CLINICAL TRIAL: NCT03893838
Title: Chromatic and Monochromatic Optical Aberrations After Corneal Refractive Surgery - Preliminary Study Assessing Their Prevalence, Methods of Reductions of Symptoms and Time-dependent Changes in Patients Symptoms
Brief Title: Chromatic and Monochromatic Optical Aberrations After Corneal Refractive Surgery
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Wrocław University of Science and Technology (Other)
Collaborators: Wroclaw Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: ST001.2018
Record Dates: First submitted 2019-03-25; First posted 2019-03-28 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Refractive Errors; Aberration, Corneal Wavefront
MeSH Terms: conditions — Refractive Errors; Corneal Wavefront Aberration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Post refractive surgery without HOA: Patients post refractive surgery that do not complain on the high order aberrations such as glare, halo and starburst.
- Post refractive surgery with HOA: Patients post refractive surgery that do complain on the high order aberrations such as glare, halo and starburst.
- Post refractive surgery with rainbow HOA: Patients post refractive surgery that do complain on:
  1. the high order aberrations such as glare, halo and starburst but with the chromatic aureola
  2. difficulties working with LCD projectors, monitors, cell phones and tablets

SUMMARY:
Refractive surgeries can be divided into two distinct categories: 1) corneal surgeries (superficial and deep procedures) carried on the surface of the eye and 2) lens surgeries (phakic IOL, refractive lens exchange) - an intraocular intervention, performed in the anterior or posterior chamber or on the lens. In the proposed protocol focus is on the corneal refractive surgeries impact on monochromatic higher-order aberrations on the one hand and chromatic aberrations on the other. During the surgery in order to get the patient emmetropic, refractive surgery corrects optical defects by decreasing aberrations of lower orders ) simultaneously increases high-order aberrations (that is perceived by the patient as halo, glare or starburst). Informations about prevalence and causes of higher order aberrations after refractive surgery are numerous but there is no information about chromatic aberrations.

ELIGIBILITY:
Inclusion Criteria:

* patient after corneal refractive surgery at least for 4 months
* post surgical refraction within +/- 0.75 diopter of spherical and +/- 1.0 diopter of cylindrical error
* willing and able to understand and sign an informed consent form.

Exclusion Criteria:

* patient unable to participate in the study
* any corneal diseases, eyes trauma or systemic diseases history; keratoconus or tendency of keratoconus
* corneal macula and obvious pannus; current enrolment in another clinical trial/research project

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients after refractive surgery
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2024-02-01 (Estimated)

PRIMARY OUTCOMES:
number of high order and chromatic aberrations after refractive surgery | 6 months
  number of high order and chromatic aberrations after refractive surgery
Chromoretinoscopy for near (MEM) and distance | 6 months
  Conducted with a modified by researchers retinoscopy with distinct filters
Aberrometry reading for corneal HOA | 6 months
  Conducted with aberrometer and corneal tomography
Transverse chromatic aberration | 6 months
  Conducted with a modified by researchers aniseikonia test (with red and green lenses)

SECONDARY OUTCOMES:
Change in Hue 100 test | 6 months
  without and after the introduction of glasses with accommodation support, a blue light filter or concave lenses up to -0,5 diopter
Change of contrast sensitivity for near vision | 6 months
  without and after the introduction of glasses with accommodation support, a blue light filter or concave lenses up to -0,5 diopter
Visual Function Questionaire 25 | 6 months
  Conducted with VFQ-25 test

CONTACTS AND LOCATIONS:
Overall Officials: Joanna Przeździecka-Dołyk, PhD, Principal Investigator — Wrocław University of Science and Technology
Locations (1):
- Department of Optics and Photonics, Wroclaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided
We intend to share anonymised data